CLINICAL TRIAL: NCT03957408
Title: An Investigational Study of Accommodation Triggering and Control to Allow for the Performance of Refraction Measurements
Brief Title: Investigational Study of Accommodation Triggering and Control to Allow for the Performance of Refraction Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeQue Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EYEQUE - 002
Record Dates: First submitted 2019-05-09; First posted 2019-05-21 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2020-01

CONDITIONS: Accommodation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visual Stimuli (Experimental): Participants will be presented various visual stimuli in which accommodative response is measured.
  Interventions: Device: Visual Stimuli

INTERVENTIONS:
Device: Visual Stimuli — Subjects will be presented various visual stimuli and may be asked to perform tasks. Their accommodative response will be measured.

SUMMARY:
An investigational study in the control of the user's accommodative state via visual stimuli.

DETAILED DESCRIPTION:
The EyeQue Corporation (EyeQue) is developing devices to measure refraction that can be used outside of the clinic. The refraction devices require the user to perform a series of tests while looking through it to view a visual display. The current devices do not currently account for accommodation and therefore may present inaccurate results for the younger population where the accommodation effect is quite significant. This study is aimed at enabling future EyeQue refraction measurement products to overcome this issue and provide the required tools to allow for accommodation measurement, correction and control. Control of the user's accommodative state will allow for measurement of near vision as well as far vision based on the refractive measurement.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 18 through 30 years at the time of consent
* Binocular vision
* Willing and able to give informed consent and follow all study procedures and requirements
* Fluent in English

Exclusion Criteria:

* Spherical correction > +4D or < -5D, astigmatism < -2.5D.
* Using anticholinergic medications (including first-generation antihistamines) or other medications known to affect visual acuity within the greater of 3 days or 5 half-lives prior to enrolling in this study
* Using an investigational drug or approved therapy for investigational use within the greater of 3 days or 5 half-lives prior to enrolling in this study
* Has initiated any new medication in the past 2 weeks that, in the best medical judgment of the investigator, would impact their participation in the study or ability to use EyeQue devices
* Reported or observed eye disease or pathology, including but not limited to:

  * Glaucoma
  * Cataracts
  * Macular degeneration
  * Eye infection
  * Keratoconus
  * Diabetic neuropathy/retinopathy
  * Cytomegalovirus retinitis
  * Color blindness (any color deficiency)
  * Diabetic macular edema
  * Amblyopia
  * Chronic or acute uveitis (cells and/or flare in anterior chamber)
  * Strabismus (exotropia, esotropia, and hypertropia)
  * Macular hole
* Eye surgery within the last 12 months (including Lasik or lens replacement)
* Subject does not have the physical dexterity to properly operate the EyeQue VisionCheck device or the EyeQue app on the smartphone in the investigator's opinion
* PD smaller than 50mm or larger than 75mm.
* Any self-reported mental illness or condition, including but not limited to: claustrophobia, fear of simulators, nyctophobia.
* Any self-reported neurological diseases, including but not limited to: epilepsy, Alzheimer's, nystagmus.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Accommodative Response | Through study completion, an average of 5 months
  Measurement of accommodative response by measuring visual refraction while the subject is viewing various visual stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Sapiens, Principal Investigator — EyeQue Corp.
Locations (1):
- EyeQue, Newark, California, United States